CLINICAL TRIAL: NCT06142032
Title: Support Groups in the Metaverse for Ukrainian Refugees: A Randomized Clinical Trial
Brief Title: Support Groups in the Metaverse for Ukrainian Refugees
Acronym: METASUPUKR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Cezar Giosan, Associate Professor of Psychology, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: METASUPPORTGROUPS
Record Dates: First submitted 2023-11-08; First posted 2023-11-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Mental Health Wellness 1; Well-Being, Psychological
Keywords: Metaverse; Refugees; Support groups; Ukraine; Mental health; Well-being; Randomized clinical trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metaverse support group (Experimental): Online intervention
  Interventions: Behavioral: Metaverse support group
- In-Person support group (Active Comparator): In-person intervention
  Interventions: Behavioral: In-Person support group
- Waitlist (No Intervention): Control

INTERVENTIONS:
Behavioral: Metaverse support group — Delivery method: Online, virtual platforms. Number of sessions: 5. Duration of each session: 1.5 hours. Sessions will adhere to evidence-based protocols for conducting support groups with a trauma-informed approach. Each session will cover a specific topic of interest related to the challenges faced by Ukrainian refugees (e.g., stress management, cultural adjustment, self-care, etc.).
  Support group session structure:
  * Introduction, check-in, ground rules;
  * Introducing the topic (topics will be chosen based on the feedback received from a previous session; the first session will cover a topic chosen by the facilitator);
  * Encouragement of participants to share thoughts, ideas and experiences;
  * Psychoeducation on the topics;
  * Summary, takeaway, feedback.
  Arms: Metaverse support group
Behavioral: In-Person support group — Delivery method: In-Person, traditional. Number of sessions: 5. Duration of each session: 1.5 hours. Sessions will adhere to evidence-based protocols for conducting support groups with a trauma-informed approach. Each session will cover a specific topic of interest related to the challenges faced by Ukrainian refugees (e.g., stress management, cultural adjustment, self-care, etc.).
  Support group session structure:
  * Introduction, check-in, ground rules;
  * Introducing the topic (topics will be chosen based on the feedback received from a previous session; the first session will cover a topic chosen by the facilitator);
  * Encouragement of participants to share thoughts, ideas and experiences;
  * Psychoeducation on the topics;
  * Summary, takeaway, feedback.
  Arms: In-Person support group

SUMMARY:
The goal of this clinical trial is to test the efficacy of support groups held in the Metaverse, designed to promote mental health and well-being in Ukrainian refugees.

Participants:

* will be allocated to one of three conditions: (1) Metaverse support group (intervention); (2) In-Person support group (intervention); or (3) Waitlist.
* will be asked to participate in 5 support group sessions, once per week, for each intervention condition.

The Metaverse support groups will be compared with the In-Person support groups and with the Waitlist, to test:

* the efficacy of the Metaverse condition compared to the In-Person condition.
* the efficacy of the intervention conditions compared to the waitlist.

DETAILED DESCRIPTION:
This protocol outlines a randomized clinical trial to assess the efficacy of virtual support groups (i.e., groups meeting in the Metaverse) for Ukrainian refugees. The study will provide essential insights into the potential benefits of using the Metaverse in delivering support group sessions. The results will contribute to the development of targeted and scalable interventions and policies to promote the well-being of Ukrainian refugees.

Participants will be recruited from Ukrainian refugee communities. The participants will be randomly assigned to one of three conditions: (1) Metaverse intervention group; (2) In-person intervention group; and (3) Waitlist. Stratification will consider factors such as age, gender, trauma history, and language proficiency to achieve balanced group distributions.

The In-Person and Metaverse groups will participate in five weekly support group sessions led by licensed psychologists.

All three groups will be evaluated at (1) pre-intervention (baseline), (2) after session no. 2, (3) post-intervention, and (4) 3-month follow-up.

G*Power analysis yields a total of N=45 (f = 0.25, power = 0.95) for the three conditions.

Statistical analysis plan: includes the analysis of primary and secondary outcomes, which will be assessed using predefined measures described at the measures section. Additionally, we will assess various predictors to gain insights into the factors influencing intervention outcomes. These predictors will be measured using specific instruments, including a screener (DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure-adult version) and Working Alliance Inventory-Short Form (WAI-S).

ELIGIBILITY:
Inclusion Criteria:

- Part of Ukrainian refugee communities

Exclusion Criteria:

* Younger than 18.
* Not part of the Ukrainian refugee community.
* Formally diagnosed with a mental disorder.
* PTSD
* Currently participating in any ongoing therapeutic intervention or treatment for mental health.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Depressive symptomatology | Up to 9 months
  Depressive symptomatology will be assessed with the Patient Health Questionnaire-Severity Measure for Depression, 9 item questionnaire. Participants assign ratings on a scale of 0 to 3 based on how often they experienced specific items in the preceding 2-week timeframe (0- not at all; 3 - nearly every day). The scores indicate the severity of depression, ranging from minimal depression (1-4) to mild, moderate, moderately severe, or severe depression (20-27).
Anxiety symptomatology | Up to 9 months
  Anxiety symptomatology will be assessed with the help of General Anxiety Disorder -7 - Severity Measure for Generalized Anxiety Disorder 7 item questionnaire.
  The measure is a 7-question self-reported instrument designed to correspond to some of the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition diagnostic criteria for GAD. Participants assign ratings on a scale of 0 to 3 based on how often they experienced specific items in the preceding 2-week timeframe (0 - not at all; 3 - nearly every day). The total score for the seven items ranges from 0 to 21(minimal anxiety, to mild, moderate and severe).

SECONDARY OUTCOMES:
Well-being | Up to 9 months
  The World Health Organization - Five Well-Being Index is used to assess the well-being of participants. The measure is a 5-item instrument consisting of statements that respondents rate on a 6-point Likert scale (0 - at no time; 5 - all of the time). The statements are rated in relation to the past two weeks. The raw scores range from 0 to 25 and are multiplied by 100 to give the final score which ranges from 0 (the worst well-being) to 100 (the best well-being).
Gender Based Violence Awareness | Up to 9 months
  Gender-based violence awareness will be assessed through five general knowledge questions about GBV. Participants will be asked to indicate the correct answer from a list of statements. Each correct answer receives one point. The total score ranges from 0 (no GBV awareness at all) to 5 (aware of GBV). The questions were developed in collaboration with an NGO focused on gender-based violence promotion among Ukrainian refugees.
Perceived Social Support | Up to 9 months
  The Multidimensional Scale of Perceived Social Support is used to assess the Perceived Social Support. The questionnaire is a 12-item self-report instrument with items measured on a 7-point Likert scale (0 - very strongly disagree; 7 - very strongly agree). Participants are asked to indicate their preference for each statement provided in the measure. The statements refer to 3 subdomains - Significant Other, Family, and Friends and the scores can be calculated both for each subscale and as a total. Total scores range from 12 to 84. Scores ranging from 12 to 35 represent low perceived social support, 36 to 60 represent medium perceived social support, and 61 to 84 represent high perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Cezar Giosan, PhD, Principal Investigator — University of Bucharest
Locations (1):
- University of Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giosan C, Popoviciu CM, Zhamaliyeva S, Zaborot I, Deac G. Evaluating the efficacy of support groups in the metaverse for Ukrainian refugees: a protocol for a randomized clinical trial. Trials. 2024 Oct 19;25(1):697. doi: 10.1186/s13063-024-08543-6. PMID 39427163